CLINICAL TRIAL: NCT01949311
Title: An Open-label Study of Dupilumab in Patients With Atopic Dermatitis Who Participated in Previous Dupilumab Clinical Trials
Brief Title: Open-label Study of Dupilumab in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1225; 2013-001449-15 (EudraCT Number)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Participants will receive repeat doses of dupilumab
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
The primary objective is to assess the long-term safety of dupilumab administered in adult participants with atopic dermatitis (AD).

The secondary objective of the study is to assess the immunogenicity of dupilumab in adult participants with AD, in the context of re-treatment, and to monitor efficacy parameters associated with long-term treatment.

Optional Sub-Study:

The primary objective of the sub-study is to assess the safety of the new dupilumab drug product in adult patients with AD after switching from the current dupilumab drug product.

The secondary objectives of the sub-study are to evaluate systemic exposure and immunogenicity of the new dupilumab drug product in adult patients with AD.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participation in a prior clinical trial of dupilumab for AD and met one of the following:

   1. Received study treatment and adequately completed the assessments required for both the treatment and follow-up periods of the parent studies (except studies listed in b) as defined in the parent protocols
   2. Received study treatment in one the studies that have completed last patient, last visit irrespective of duration of participation, provided that patients completed with the instructions received during the study.
   3. Underwent screening in R668-AD-1334 (Liberty AD SOLO 1) or R668-AD-1416 (Liberty AD SOLO 2) but could not be randomized due to randomization closure.
2. Willing and able to comply with all clinic visits and study-related procedures
3. Able to understand and complete study-related questionnaires
4. Provide signed informed consent

Optional Sub-Study:

1. Provide separate informed consent
2. Continuing in the treatment period of the main OLE study
3. Demonstrated compliance with dupilumab therapy, as defined in the protocol

Key Exclusion Criteria:

1. Patients who, during their participation in a previous dupilumab clinical trial, developed a serious adverse event (SAE) deemed related to dupilumab*, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with dupilumab may present an unreasonable risk for the patient.
2. Patients who, during their participation in a previous dupilumab clinical trial, developed an AE that was deemed related to dupilumab* and led to study treatment discontinuation, which in the opinion of the investigator or of the medical monitor could indicate that continued treatment with dupilumab may present an unreasonable risk for the patient.
3. Conditions in the previous dupilumab study consistent with protocol-defined criteria for permanent study drug discontinuation, if deemed related to dupilumab* or led to investigator - or sponsor-initiated withdrawal of patient from the study (eg, non-compliance, inability to complete study assessments, etc.).

   *Note for exclusion criteria # 1, 2, and 3: In studies that are still blinded, conditions deemed related to the study treatment will be considered related to dupilumab.
4. Treatment with an investigational drug, other than dupilumab, within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
5. Pregnant or breastfeeding women, or planning to become pregnant or breastfeed during the patient's participation in this study

Optional Sub-Study:

1. Patients who have already completed the end of treatment visit (ie, visit 44) for the main study R668-AD-1225

Note: Other Protocol Defined Inclusion / Exclusion Criteria Apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2733 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (418):
- United States (115):
  - Regeneron Study Site, Anniston, Alabama
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site 1, Birmingham, Alabama
  - Regeneron Study Site 2, Birmingham, Alabama
  - Regeneron Study Site 2, Phoenix, Arizona
  - Regeneron Study Site 3, Phoenix, Arizona
  - Regeneron Study Site 1, Phoenix, Arizona
  - Regeneron Study Site, Fort Smith, Arkansas
  - Regeneron Study Site, Rogers, Arkansas
  - Regeneron Study Site, Bakersfield, California
  - Regeneron Study Site, Clovis, California
  - Regeneron Study Site, Costa Mesa, California
  - Regeneron Study Site, Encinitas, California
  - Regeneron Study Site, Fremont, California
  - Regeneron Study Site, Lomita, California
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site 1, Los Angeles, California
  - Regeneron Study Site 2, Los Angeles, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Oceanside, California
  - Regeneron Study Site, Orange, California
  - Regeneron Study Site, Rolling Hills Estates, California
  - Regeneron Study Site, San Diego, California
  - Regeneron Study Site 1, San Diego, California
  - Regeneron Study Site 2, San Diego, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Centennial, Colorado
  - Regeneron Study Site, Denver, Colorado
  - Regeneron Study Site, Trumbull, Connecticut
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Boca Raton, Florida
  - Regeneron Study Site, Clearwater, Florida
  - Regeneron Study Site, Fort Lauderdale, Florida
  - Regeneron Study Site 1, Jacksonville, Florida
  - Regeneron Study Site 2, Jacksonville, Florida
  - Regeneron Study Site, Lake Worth, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Miami Lakes, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, West Palm Beach, Florida
  - Regeneron Study Site, Alpharetta, Georgia
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Columbus, Georgia
  - Regeneron Study Site, Macon, Georgia
  - Regeneron Study Site, Newnan, Georgia
  - Regeneron Study Site, Sandy Springs, Georgia
  - Regeneron Study Site, Savannah, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Normal, Illinois
  - Regeneron Study Site, West Dundee, Illinois
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Newburgh, Indiana
  - Regeneron Study Site, Plainfield, Indiana
  - Regeneron Study Site, Overland Park, Kansas
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Rockville, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Bay City, Michigan
  - Regeneron Study Site, Farmington Hills, Michigan
  - Regeneron Study Site, Troy, Michigan
  - Regeneron Study Site, Edina, Minnesota
  - Regeneron Study Site, Fridley, Minnesota
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Plymouth, Minnesota
  - Regeneron Study Site, Saint Joseph, Missouri
  - Regeneron Study Site, St Louis, Missouri
  - Regeneron Study Site, Henderson, Nevada
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Portsmouth, New Hampshire
  - Regeneron Study Site, Berlin, New Jersey
  - Regeneron Study Site, East Windsor, New Jersey
  - Regeneron Study Site, Verona, New Jersey
  - Regeneron Study Site 1, Albuquerque, New Mexico
  - Regeneron Study Site 2, Albuquerque, New Mexico
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site, Corning, New York
  - Regeneron Study Site, Forest Hills, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Rochester, New York
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, High Point, North Carolina
  - Regeneron Study Site, Raleigh, North Carolina
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Winston-Salem, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Norman, Oklahoma
  - Regeneron Study Site, Tulsa, Oklahoma
  - Regeneron Study Site, Medford, Oregon
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Bethlehem, Pennsylvania
  - Regeneron Study Site, Jenkintown, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Pittsburgh, Pennsylvania
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Greer, South Carolina
  - Regeneron Study Site, Chattanooga, Tennessee
  - Regeneron Study Site, Nashville, Tennessee
  - Regeneron Study Site, Arlington, Texas
  - Regeneron Study Site, Austin, Texas
  - Regeneron Study Site, Bellaire, Texas
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site 1, San Antonio, Texas
  - Regeneron Study Site 2, San Antonio, Texas
  - Regeneron Study Site, Waco, Texas
  - Regeneron Study Site, Webster, Texas
  - Regeneron Study Site, Salt Lake City, Utah
  - Regeneron Study Site, South Burlington, Vermont
  - Regeneron Study Site, Newport News, Virginia
  - Regeneron Study Site, Norfolk, Virginia
  - Regeneron Study Site, Richmond, Virginia
  - Regeneron Study Site, Seattle, Washington
- Australia (8):
  - Regeneron Study Site, Phillip, Australian Capital Territory
  - Regeneron Study Site, Kogarah, New South Wales
  - Regeneron Study Site, Benowa, Queensland
  - Regeneron Study Site, Woolloongabba, Queensland
  - Regeneron Study Site, Hectorville, South Australia
  - Regeneron Study Site, Carlton, Victoria
  - Regeneron Study Site, East Melbourne, Victoria
  - Regeneron Study Site, Fremantle, Western Australia
- Austria (2):
  - Regeneron Study Site 1, Vienna
  - Regeneron Study Site 2, Vienna
- Belgium (3):
  - Regeneron Study Site, Brussels, Brussels Capital
  - Regeneron Study Site, Loverval, Hainaut
  - Regeneron Study Site, Leuven, Vlaams Brabant
- Bulgaria (3):
  - Regeneron Study Site, Dupnitsa, Kyustendil
  - Regeneron Study Site 1, Sofia, Sofia-Grad
  - Regeneron Study Site 2, Sofia, Sofia-Grad
- Canada (36):
  - Regeneron Study Site 1, Calgary, Alberta
  - Regeneron Study Site 2, Calgary, Alberta
  - Regeneron Study Site 1, Edmonton, Alberta
  - Regeneron Study Site 2, Edmonton, Alberta
  - Regeneron Study Site 1, Surrey, British Columbia
  - Regeneron Study Site 2, Surrey, British Columbia
  - Regeneron Study Site 1, Vancouver, British Columbia
  - Regeneron Study Site 2, Vancouver, British Columbia
  - Regeneron Study Site 3, Vancouver, British Columbia
  - Regeneron Study Site 1, Winnipeg, Manitoba
  - Regeneron Study Site, Bathurst, New Brunswick
  - Regeneron Study Site, St. John's, Newfoundland and Labrador
  - Regeneron Study Site, Ajax, Ontario
  - Regeneron Study Site 1, Barrie, Ontario
  - Regeneron Study Site 2, Barrie, Ontario
  - Regeneron Study Site, Etobicoke, Ontario
  - Regeneron Study Site 1, Hamilton, Ontario
  - Regeneron Study Site 2, Hamilton, Ontario
  - Regeneron Study Site, Markham, Ontario
  - Regeneron Study Site, Mississauga, Ontario
  - Regeneron Study Site, Newmarket, Ontario
  - Regeneron Study Site, North Bay, Ontario
  - Regeneron Study Site, Oakville, Ontario
  - Regeneron Study Site 1, Ottawa, Ontario
  - Regeneron Study Site, Peterborough, Ontario
  - Regeneron Study Site 1, Richmond Hill, Ontario
  - Regeneron Study Site 2, Richmond Hill, Ontario
  - Regeneron Study Site, Toronto, Ontario
  - Regeneron Study Site, Waterloo, Ontario
  - Regeneron Study Site 1, Windsor, Ontario
  - Regeneron Study Site 2, Windsor, Ontario
  - Regeneron Study Site, Drummondville, Quebec
  - Regeneron Study Site, Montreal, Quebec
  - Regeneron Study Site 3, Ste-Foy, Quebec
  - Regeneron Study Site, Ste-Foy
  - Regeneron Study Site, Winnipeg
- Regeneron Study Site, Hong Kong, China
- Czechia (6):
  - Regeneron Study Site, Hradec Králové
  - Regeneron Study Site, Kutná Hora
  - Regeneron Study Site, Náchod
  - Regeneron Study Site, Prague
  - Regeneron Study Site, Svitavy
  - Regeneron Study Site, Ústí nad Labem
- Denmark (4):
  - Regeneron Study Site, Copenhagen, Capital
  - Regeneron Study Site, Hellerup, Capital
  - Regeneron Study Site, Aarhus, Central Jutland
  - Regeneron Study Site, Roskilde, Zeeland
- Estonia (5):
  - Regeneron Study Site 1, Tallinn, Harju
  - Regeneron Study Site 2, Tallinn, Harju
  - Regeneron Study Site 3, Tallinn, Harju
  - Regeneron Study Site 1, Tartu, Tartu
  - Regeneron Study Site 2, Tartu, Tartu
- Finland (3):
  - Regeneron Study Site, Helsinki, Etelä-Suomen Iääni
  - Regeneron Study Site, Turku, Etelä-Suomen Lääni
  - Regeneron Study Site, Tampere, Länsi-Suomen Lääni
- France (8):
  - Regeneron Study Site, Nice, Alpes-Maritimes
  - Regeneron Study Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Regeneron Study Site, Marseille, Bouches-du-Rhône
  - Regeneron Study Site, Reims, Marne
  - Regeneron Study Site, Lille, Nord
  - Regeneron Study Site, Lille
  - Regeneron Study Site, Nantes
  - Regeneron Study Site, Paris, Île-de-France Region
- Germany (44):
  - Regeneron Study Site, Friedrichshafen, Baden-Wurttemberg
  - Regeneron Study Site, Heidelberg, Baden-Wurttemberg
  - Regeneron Study Site, Langenau, Baden-Wurttemberg
  - Regeneron Study Site, Stuttgart, Baden-Wurttemberg
  - Regeneron Study Site, Tübingen, Baden-Wurttemberg
  - Regeneron Study Site, Augsburg, Bavaria
  - Regeneron Study Site, Erlangen, Bavaria
  - Regeneron Study Site, Munich, Bavaria
  - Regeneron Study Site, München, Bavaria
  - Regeneron Study Site, Mahlow, Brandenburg
  - Regeneron Study Site 2, Hamburg, Hamburg
  - Regeneron Study Site, Frankfurt am Main, Hesse
  - Regeneron Study Site, Hanover, Lower Saxony
  - Regeneron Study Site, Schwerin, Mecklenburg-Vorpommern
  - Regeneron Study Site 1, Bochum, North Rhine-Westphalia
  - Regeneron Study Site 2, Bochum, North Rhine-Westphalia
  - Regeneron Study Site, Dülmen, North Rhine-Westphalia
  - Regeneron Study Site, Ibbenbueren, North Rhine-Westphalia
  - Regeneron Study Site, Mönchengladbach, North Rhine-Westphalia
  - Regeneron Study Site, Münster, North Rhine-Westphalia
  - Regeneron Study Site, Mainz, Rhineland-Palatinate
  - Regeneron Study Site, Selters, Rhineland-Palatinate
  - Regeneron Study Site 1, Dresden, Saxony
  - Regeneron Study Site 2, Dresden, Saxony
  - Regeneron Study Site 3, Dresden, Saxony
  - Regeneron Study Site, Leipzig, Saxony
  - Regeneron Study Site, Halle, Saxony-Anhalt
  - Regeneron Study Site, Magdeburg, Saxony-Anhalt
  - Regeneron Study Site 1, Kiel, Schleswig-Holstein
  - Regeneron Study Site 2, Kiel, Schleswig-Holstein
  - Regeneron Study Site, Lübeck, Schleswig-Holstein
  - Regeneron Study Site, Gera, Thuringia
  - Regeneron Study Site 1, Berlin
  - Regeneron Study Site 2, Berlin
  - Regeneron Study Site 3, Berlin
  - Regeneron Study Site 4, Berlin
  - Regeneron Study Site 5, Berlin
  - Regeneron Study Site 6, Berlin
  - Regeneron Study Site 7, Berlin
  - Regeneron Study Site, Bonn
  - Regeneron Study Site, Darmstadt
  - Regeneron Study Site 1, Hamburg
  - Regeneron Study Site, Münster
  - Regeneron Study Site, Osnabrück
- Hungary (9):
  - Regeneron Study Site, Orosháza, Bekes County
  - Regeneron Study Site, Sátoraljaújhely, Borsod-Abauj Zemplen county
  - Regeneron Study Site, Szeged, Csongrád megye
  - Regeneron Study Site, Szolnok, Jász-Nagykun-Szolnok
  - Regeneron Study Site, Kaposvár, Somogy County
  - Regeneron Study Site 1, Budapest
  - Regeneron Study Site 2, Budapest
  - Regeneron Study Site 3, Budapest
  - Regeneron Study Site, Veszprém
- Regeneron Study Site, Dublin, Ireland
- Italy (14):
  - Regeneron Study Site, Bologna, Balogna
  - Regeneron Study Site, Ancona
  - Regeneron Study Site, Chieti
  - Regeneron Study Site, Florence
  - Regeneron Study Site, Lucca
  - Regeneron Study Site, L’Aquila
  - Regeneron Study Site, Messina
  - Regeneron Study Site, Milan
  - Regeneron Study Site, Novara
  - Regeneron Study Site, Pavia
  - Regeneron Study Site, Perugia
  - Regeneron Study Site, Pisa
  - Regeneron Study Site 1, Roma
  - Regeneron Study Site 2, Roma
- Japan (59):
  - Regeneron Study Site, Nagakute, Aichi-ken
  - Regeneron Study Site, Kurume, Fukuoka
  - Regeneron Study Site, Fukuyama, Hiroshima
  - Regeneron Study Site, Sapporo, Hokkaido
  - Regeneron Study Site 1, Fukuoka, Hukuoka
  - Regeneron Study Site 2, Fukuoka, Hukuoka
  - Regeneron Study Site, Kitakyushu, Hukuoka
  - Regeneron Study Site 1, Amagasaki, Hyôgo
  - Regeneron Study Site 2, Amagasaki, Hyôgo
  - Regeneron Study Site, Inashiki-gun, Ibaraki
  - Regeneron Study Site 1, Yokohama, Kanagawa
  - Regeneron Study Site 2, Yokohama, Kanagawa
  - Regeneron Study Site 3, Yokohama, Kanagawa
  - Regeneron Study Site, Kamimashiki, Kumamoto
  - Regeneron Study Site, Habikino, Osaka
  - Regeneron Study Site, Neyagawa, Osaka
  - Regeneron Study Site, Sakai, Osaka
  - Regeneron Study Site, Takatsuki, Osaka
  - Regeneron Study Site, Hamamatsu, Shizuoka
  - Regeneron Study Site, Yaizu, Shizuoka
  - Regeneron Study Site 1, Bunkyo-ku, Tokyo
  - Regeneron Study Site 2, Bunkyo-ku, Tokyo
  - Regeneron Study Site 1, Chiyoda-ku, Tokyo
  - Regeneron Study Site 2, Chiyoda-ku, Tokyo
  - Regeneron Study Site, Chuo-ku, Tokyo
  - Regeneron Study Site, Koto-ku, Tokyo
  - Regeneron Study Site, Nakano-ku, Tokyo
  - Regeneron Study Site 1, Nerima City, Tokyo
  - Regeneron Study Site 2, Nerima City, Tokyo
  - Regeneron Study Site, Ōta-ku, Tokyo
  - Regeneron Study Site, Setagaya-ku, Tokyo
  - Regeneron Study Site 1, Shibuya-ku, Tokyo
  - Regeneron Study Site 2, Shibuya-ku, Tokyo
  - Regeneron Study Site 3, Shibuya-ku, Tokyo
  - Regeneron Study Site 1, Shinagawa-ku, Tokyo
  - Regeneron Study Site 2, Shinagawa-ku, Tokyo
  - Regeneron Study Site 1, Shinjuku-ku, Tokyo
  - Regeneron Study Site 2, Shinjuku-ku, Tokyo
  - Regeneron Study Site 3, Shinjuku-ku, Tokyo
  - Regeneron Study Site 4, Shinjuku-ku, Tokyo
  - Regeneron Study Site 5, Shinjuku-ku, Tokyo
  - Regeneron Study Site 6, Shinjuku-ku, Tokyo
  - Regeneron Study Site 1, Suginami, Tokyo
  - Regeneron Study Site 2, Suginami, Tokyo
  - Regeneron Study Site, Chūō, Yamanashi
  - Regeneron Study Site, Kofu, Yamanashi
  - Regeneron Study Site 2, Fukuyama
  - Regeneron Study Site, Gifu
  - Regeneron Study Site 1, Hiroshima
  - Regeneron Study Site 2, Hiroshima
  - Regeneron Study Site 1, Kyoto
  - Regeneron Study Site 2, Kyoto
  - Regeneron Study Site 1, Osaka
  - Regeneron Study Site 2, Osaka
  - Regeneron Study Site, Saitama
  - Regeneron Study Site 3, Shinagawa-ku
  - Regeneron Study Site, Suginome
  - Regeneron Study Site, Wakayama
  - Regeneron Study Site 4, Yokohama
- Lithuania (5):
  - Regeneron Study Site, Kaunas, Kaunas County
  - Regeneron Study Site 1, Vilnius, Vilnius County
  - Regeneron Study Site 2, Vilnius, Vilnius County
  - Regeneron Study Site 1, Klaipėda
  - Regeneron Study Site 2, Klaipėda
- Netherlands (5):
  - Regeneron Study Site, Breda, North Brabant
  - Regeneron Study Site, Amsterdam, North Holland
  - Regeneron Study Site, Rotterdam, South Holland
  - Regeneron Study Site, Groningen
  - Regeneron Study Site, Utrecht
- New Zealand (2):
  - Regeneron Study Site, Dunedin, South Island
  - Regeneron Study Site, Auckland
- Poland (36):
  - Regeneron Study Site 1, Poznan, Greater Poland Voivodeship
  - Regeneron Study Site 2, Poznan, Greater Poland Voivodeship
  - Regeneron Study Site 3, Poznan, Greater Poland Voivodeship
  - Regeneron Study Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Regeneron Study Site 1, Krakow, Lesser Poland Voivodeship
  - Regeneron Study Site 2, Krakow, Lesser Poland Voivodeship
  - Regeneron Study Site 3, Krakow, Lesser Poland Voivodeship
  - Regeneron Study Site 1, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Study Site 2, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Study Site 3, Wroclaw, Lower Silesian Voivodeship
  - Regeneron Study Site, Lublin, Lublin Voivodeship
  - Regeneron Study Site 1, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 2, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 3, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 4, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 5, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 6, Warsaw, Masovian Voivodeship
  - Regeneron Study Site 7, Warsaw, Masovian Voivodeship
  - Regeneron Study Site, Strzelce Opolskie, Opole Voivodeship
  - Regeneron Study Site, Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Regeneron Study Site 1, Gdansk, Pomeranian Voivodeship
  - Regeneron Study Site 2, Gdansk, Pomeranian Voivodeship
  - Regeneron Study Site, Szczecin, West Pomeranian Voivodeship
  - Regeneron Study Site, Bialystok
  - Regeneron Study Site, Bydgoszcz
  - Regeneron Study Site, Chorzów
  - Regeneron Study Site, Elblag
  - Regeneron Study Site 1, Katowice
  - Regeneron Study Site 2, Katowice
  - Regeneron Study Site 3, Katowice
  - Regeneron Study Site, Ostrowiec Świętokrzyski
  - Regeneron Study Site, Skarżysko-Kamienna
  - Regeneron Study Site, Zgierz
  - Regeneron Study Site 1, Lodz, Łódź Voivodeship
  - Regeneron Study Site 2, Lodz, Łódź Voivodeship
  - Regeneron Study Site 3, Lodz, Łódź Voivodeship
- Regeneron Study Site, Brasov, Romania
- Russia (5):
  - Regeneron Study Site, Moscow, Koskva
  - Regeneron Study Site, Ryazan, Ryazan Oblast
  - Regeneron Study Site, Saint Petersburg, Sankt-Peterburg
  - Regeneron Study Site, Kazan', Tatarstan Respublika
  - Regeneron Study Site, Chelyabinsk
- Singapore (3):
  - Regeneron Study Site 1, Singapore, Central Singapore
  - Regeneron Study Site 2, Singapore, Central Singapore
  - Regeneron Study Site, Singapore, South West
- Slovakia (2):
  - Regeneron Study Site, Košice
  - Regeneron Study Site, Svidník
- South Korea (15):
  - Regeneron Study Site, Busan, Busan Gwang'yeogsi
  - Regeneron Study Site, Bucheon-si, Kyonggi-do
  - Regeneron Study Site, Hwaseong-si, Kyonggi-do
  - Regeneron Study Site, Suwon, Kyonggi-do
  - Regeneron Study Site, Uijeongbu-si, Kyonggi-do
  - Regeneron Study Site 1, Incheon
  - Regeneron Study Site 2, Incheon
  - Regeneron Study Site 1, Seoul
  - Regeneron Study Site 2, Seoul
  - Regeneron Study Site 3, Seoul
  - Regeneron Study Site 4, Seoul
  - Regeneron Study Site 5, Seoul
  - Regeneron Study Site 6, Seoul
  - Regeneron Study Site 7, Seoul
  - Regeneron Study Site 8, Seoul
- Spain (10):
  - Regeneron Study Site, Elche, Alicante
  - Regeneron Study Site, Badalona, Barcelona
  - Regeneron Study Site, Las Palmas de Gran Canaria, Canary Islands
  - Regeneron Study Site 1, Barcelona
  - Regeneron Study Site 2, Barcelona
  - Regeneron Study Site 3, Barcelona
  - Regeneron Study Site 4, Barcelona
  - Regeneron Study Site 1, Madrid
  - Regeneron Study Site 2, Madrid
  - Regeneron Study Site, Seville
- United Kingdom (13):
  - Regeneron Study Site, Dundee, Angus
  - Regeneron Study Site, Edgbaston, Birmingham
  - Regeneron Study Site, Plymouth, Devon
  - Regeneron Study Site, Portsmouth, Hampshire
  - Regeneron Study Site, Sidcup, Kent
  - Regeneron Study Site, Northwood, London
  - Regeneron Study Site, Oxford, Oxfordshire
  - Regeneron Study Site, Liverpool
  - Regeneron Study Site 1, London
  - Regeneron Study Site 2, London
  - Regeneron Study Site, Manchester
  - Regeneron Study Site, Salford
  - Regeneron Study Site, Sheffield

REFERENCES:
- [Derived] Simpson EL, Bissonnette R, Deleuran M, Nakahara T, Galus R, de Bruin-Weller M, Coleman A, van Spall M, Chen Z, Avetisova E, Bastian M, Khokhar FA. Dupilumab Treatment Up to 5 Years Shows No Clinically Meaningful Changes in Laboratory Parameters in Adults with Moderate-to-Severe Atopic Dermatitis. Adv Ther. 2026 Jan 21. doi: 10.1007/s12325-025-03458-3. Online ahead of print. PMID 41563707
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Blauvelt A, Wollenberg A, Eichenfield LF, Zhang H, Sierka D, Khokhar FA, Vakil J, Shabbir A, Marco AR, Cyr SL. No Increased Risk of Overall Infection in Adults with Moderate-to-Severe Atopic Dermatitis Treated for up to 4 Years with Dupilumab. Adv Ther. 2023 Jan;40(1):367-380. doi: 10.1007/s12325-022-02322-y. Epub 2022 Nov 1. PMID 36318387
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Beck LA, Deleuran M, Bissonnette R, de Bruin-Weller M, Galus R, Nakahara T, Seo SJ, Khokhar FA, Vakil J, Xiao J, Marco AR, Levit NA, O'Malley JT, Shabbir A. Dupilumab Provides Acceptable Safety and Sustained Efficacy for up to 4 Years in an Open-Label Study of Adults with Moderate-to-Severe Atopic Dermatitis. Am J Clin Dermatol. 2022 May;23(3):393-408. doi: 10.1007/s40257-022-00685-0. Epub 2022 May 3. PMID 35503163
- [Derived] Armstrong A, Blauvelt A, Simpson EL, Smith CH, Herranz P, Kataoka Y, Seo SJ, Ferrucci SM, Chao J, Chen Z, Rossi AB, Shumel B, Tomondy P. Continued Treatment with Dupilumab is Associated with Improved Efficacy in Adults with Moderate-to-Severe Atopic Dermatitis Not Achieving Optimal Responses with Short-Term Treatment. Dermatol Ther (Heidelb). 2022 Jan;12(1):195-202. doi: 10.1007/s13555-021-00643-4. Epub 2021 Dec 13. PMID 34897582
- [Derived] Yosipovitch G, de Bruin-Weller M, Armstrong A, Wu JJ, Herranz P, Thaci D, Delevry D, Bagousse GB, Zhang R, Shumel B, Rossi AB, Chao J. Dupilumab Treatment Provides Sustained Improvements Over 2 Years in Symptoms and Quality of Life in Adults with Atopic Dermatitis. Dermatol Ther (Heidelb). 2021 Dec;11(6):2147-2157. doi: 10.1007/s13555-021-00630-9. Epub 2021 Oct 29. PMID 34714527
- [Derived] Beck LA, Thaci D, Deleuran M, de Bruin-Weller M, Chen Z, Khokhar FA, Zhang M, Ozturk ZE, Shumel B. Laboratory safety of dupilumab for up to 3 years in adults with moderate-to-severe atopic dermatitis: results from an open-label extension study. J Dermatolog Treat. 2022 May;33(3):1608-1616. doi: 10.1080/09546634.2020.1871463. Epub 2021 Feb 8. PMID 33557637
- [Derived] Beck LA, Thaci D, Deleuran M, Blauvelt A, Bissonnette R, de Bruin-Weller M, Hide M, Sher L, Hussain I, Chen Z, Khokhar FA, Beazley B, Ruddy M, Patel N, Graham NMH, Ardeleanu M, Shumel B. Dupilumab Provides Favorable Safety and Sustained Efficacy for up to 3 Years in an Open-Label Study of Adults with Moderate-to-Severe Atopic Dermatitis. Am J Clin Dermatol. 2020 Aug;21(4):567-577. doi: 10.1007/s40257-020-00527-x. PMID 32557382

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1297 participants completed the study and 1380 participants had withdrawn. Withdrawal from study included study terminated by the Sponsor (708), and withdrawal by the participant (375), Adverse Event (107), Lost to Follow-Up (73), Lack of Efficacy (50), Protocol Deviation (34), Pregnancy (20), Physician Decision (9), and reasons not specified (4)
Groups:
- Dupilumab: Participants received repeated doses of dupilumab
Period: Overall Study
Arm/Group | Dupilumab
Started | 2677
Completed | 1297
Not Completed | 1380
Not completed — Lost to Follow-up | 73
Not completed — Terminated by Sponsor | 708
Not completed — Withdrawal by Subject | 375
Not completed — Lack of Efficacy | 50
Not completed — Protocol Deviation | 34
Not completed — Pregnancy | 20
Not completed — Physician Decision | 9
Not completed — Other | 4
Not completed — Adverse Event | 107

BASELINE CHARACTERISTICS:
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1066
  Male | 1611
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 94
  Not Hispanic or Latino | 2532
  Unknown or Not Reported | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 541
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 147
  White | 1936
  More than one race | 33
  Unknown or Not Reported | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Up to 272 weeks
Population: The safety analysis set (SAF) will include all patients who received any study drug; it is based on the treatment received (as treated).
Measure: Number; unit: Number of Events
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Number of Events | 14717

2. Primary Outcome: OPTIONAL SUB-STUDY: Number of Adverse Events of Special Interest (AESIs) Through the Last Study Visit After Switching to the New Dupilumab Drug Product
Description: Adverse events of special interest in this study include: Anaphylactic reactions, Systemic hypersensitivity reactions, Helminthic infections, Any severe type of conjunctivitis or blepharitis, Keratitis, Clinically symptomatic eosinophilia (or eosinophilia associated with clinical symptoms)
Time Frame: Up to 24 Weeks
Population: The sub-study SAF includes all patients who receive new dupilumab drug product in the sub-study.
Measure: Number; unit: Events
Groups:
- Dupilumab: Participants received repeated doses of dupilumab during the Ophthalmology Sub-study
Arm/Group | Dupilumab
Number analyzed (Participants) | 50
Events | 0

3. Secondary Outcome: Number of Serious Adverse Events (SAEs) of Special Interest
Description: as for outcome 2
Time Frame: Up to 272 weeks
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Events | 9

4. Secondary Outcome: Rate of AESIs
Description: Rate (events per patient-year) of AESIs
  Adverse events of special interest in this study include: Anaphylactic reactions, Systemic hypersensitivity reactions, Helminthic infections, Any severe type of conjunctivitis or blepharitis, Keratitis, Clinically symptomatic eosinophilia (or eosinophilia associated with clinical symptoms)
Time Frame: Up to 272 weeks
Population: as for outcome 1
Measure: Number; unit: Events per Patient-Year
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Events per Patient-Year | 2.762

5. Secondary Outcome: Number of AESIs
Description: as for outcome 2
Time Frame: Up to 272 weeks
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Events | 161

6. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score = 0-1 at Each Visit
Description: IGA is an assessment scale used to determine severity of hand and foot AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration.
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 4, 16, 36, 52, 100, 124, 156, 172, 188, 204, 220, 236, 272 (End of Study)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Baseline of study | 12.0
  Week 4: number analyzed (Participants) | 2650
  Week 4 | 31.1
  Week 16: number analyzed (Participants) | 2590
  Week 16 | 46.7
  Week 36: number analyzed (Participants) | 1313
  Week 36 | 46.2
  Week 52: number analyzed (Participants) | 893
  Week 52 | 53.8
  Week 100: number analyzed (Participants) | 1019
  Week 100 | 58.2
  Week 124: number analyzed (Participants) | 478
  Week 124 | 59.6
  Week 156: number analyzed (Participants) | 116
  Week 156 | 67.2
  Week 172: number analyzed (Participants) | 187
  Week 172 | 71.1
  Week 188: number analyzed (Participants) | 62
  Week 188 | 56.5
  Week 204: number analyzed (Participants) | 101
  Week 204 | 64.4
  Week 220: number analyzed (Participants) | 138
  Week 220 | 81.2
  Week 236: number analyzed (Participants) | 10
  Week 236 | 50.0
  End of Study (Extension): number analyzed (Participants) | 326
  End of Study (Extension) | 67.5

7. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index (EASI)-75 (≥75% Reduction in EASI Scores From Baseline of the Parent Study) at Each Visit
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 4, 16, 36, 52, 100, 124, 156, 172, 188, 204, 220, 236, 272 (End of Study)"
Population: The safety analysis set (SAF) will include all patients who received any study drug; it is based on the treatment received (as treated). Here 'n' = number of evaluable participants at the specified timeframe
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Baseline of study: number analyzed (Participants) | 2647
  Baseline of study | 33.4
  Week 4: number analyzed (Participants) | 2620
  Week 4 | 65.3
  Week 16: number analyzed (Participants) | 2560
  Week 16 | 82.0
  Week 36: number analyzed (Participants) | 1289
  Week 36 | 85.3
  Week 52: number analyzed (Participants) | 883
  Week 52 | 88.8
  Week 100: number analyzed (Participants) | 999
  Week 100 | 91.4
  Week 124: number analyzed (Participants) | 473
  Week 124 | 92.0
  Week 156: number analyzed (Participants) | 114
  Week 156 | 89.5
  Week 172: number analyzed (Participants) | 187
  Week 172 | 94.1
  Week 188: number analyzed (Participants) | 62
  Week 188 | 96.8
  Week 204: number analyzed (Participants) | 99
  Week 204 | 90.9
  Week 220: number analyzed (Participants) | 138
  Week 220 | 93.5
  Week 236: number analyzed (Participants) | 10
  Week 236 | 100
  End of Study (Extension): number analyzed (Participants) | 324
  End of Study (Extension) | 88.9

8. Secondary Outcome: Percentage of Participants With Low Disease Activity State (eg, IGA ≤2) at Each Visit
Description: Low disease activity state is defined as an IGA score of ≤2 [mild = 2, almost clear = 1, or clear = 0]
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Baseline of study | 34.7
  Week 4: number analyzed (Participants) | 2650
  Week 4 | 70.0
  Week 16: number analyzed (Participants) | 2590
  Week 16 | 83.0
  Week 36: number analyzed (Participants) | 1313
  Week 36 | 84.6
  Week 52: number analyzed (Participants) | 893
  Week 52 | 89.6
  Week 100: number analyzed (Participants) | 1019
  Week 100 | 90.9
  Week 124: number analyzed (Participants) | 478
  Week 124 | 93.1
  Week 156: number analyzed (Participants) | 116
  Week 156 | 94.8
  Week 172: number analyzed (Participants) | 187
  Week 172 | 96.3
  Week 188: number analyzed (Participants) | 62
  Week 188 | 96.8
  Week 204: number analyzed (Participants) | 101
  Week 204 | 96.0
  Week 220: number analyzed (Participants) | 138
  Week 220 | 97.1
  Week 236: number analyzed (Participants) | 10
  Week 236 | 90.0
  End of Study (Extension): number analyzed (Participants) | 326
  End of Study (Extension) | 92.6

9. Secondary Outcome: Change From Baseline in EASI Score at Each Visit
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Score on a scale
  Week 4: number analyzed (Participants) | 2650
  Week 4 | -8.59 (10.196)
  Week 16: number analyzed (Participants) | 2590
  Week 16 | -11.89 (12.583)
  Week 36: number analyzed (Participants) | 1313
  Week 36 | -17.32 (13.989)
  Week 52: number analyzed (Participants) | 894
  Week 52 | -16.46 (13.719)
  Week 100: number analyzed (Participants) | 1019
  Week 100 | -17.99 (14.049)
  Week 124: number analyzed (Participants) | 478
  Week 124 | -17.68 (13.794)
  Week 156: number analyzed (Participants) | 116
  Week 156 | -14.23 (14.358)
  Week 172: number analyzed (Participants) | 187
  Week 172 | -13.23 (13.651)
  Week 188: number analyzed (Participants) | 62
  Week 188 | -19.24 (11.253)
  Week 204: number analyzed (Participants) | 101
  Week 204 | -14.50 (15.615)
  Week 220: number analyzed (Participants) | 138
  Week 220 | -12.75 (14.444)
  Week 236: number analyzed (Participants) | 10
  Week 236 | -16.69 (9.743)
  End of Study (Extension): number analyzed (Participants) | 326
  End of Study (Extension) | -13.14 (14.614)

10. Secondary Outcome: Percent Change From Baseline in EASI Score at Each Visit
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percent of Change
  Week 4: number analyzed (Participants) | 2584
  Week 4 | -42.02 (88.963)
  Week 16: number analyzed (Participants) | 2527
  Week 16 | -54.82 (316.630)
  Week 36: number analyzed (Participants) | 1304
  Week 36 | -60.40 (603.886)
  Week 52: number analyzed (Participants) | 885
  Week 52 | -75.76 (73.014)
  Week 100: number analyzed (Participants) | 1013
  Week 100 | -82.61 (29.534)
  Week 124: number analyzed (Participants) | 477
  Week 124 | -84.15 (27.737)
  Week 156: number analyzed (Participants) | 115
  Week 156 | -83.45 (32.410)
  Week 172: number analyzed (Participants) | 178
  Week 172 | -74.98 (78.138)
  Week 188: number analyzed (Participants) | 62
  Week 188 | -88.72 (15.122)
  Week 204: number analyzed (Participants) | 101
  Week 204 | -70.91 (74.941)
  Week 220: number analyzed (Participants) | 129
  Week 220 | -30.79 (370.994)
  Week 236: number analyzed (Participants) | 10
  Week 236 | -87.56 (10.851)
  End of Study (Extension): number analyzed (Participants) | 316
  End of Study (Extension) | -55.44 (213.819)

11. Secondary Outcome: Percentage of Participants With EASI-50 (≥50% Reduction in EASI Scores From Baseline of the Parent Study) at Each Visit
Description: EASI-50 was defined as >=50% reduction in EASI scores from baseline of the parent study
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Week 4: number analyzed (Participants) | 2620
  Week 4 | 86.0
  Week 16: number analyzed (Participants) | 2560
  Week 16 | 95.0
  Week 36: number analyzed (Participants) | 1289
  Week 36 | 96.7
  Week 52: number analyzed (Participants) | 883
  Week 52 | 97.4
  Week 100: number analyzed (Participants) | 999
  Week 100 | 98.5
  Week 124: number analyzed (Participants) | 473
  Week 124 | 98.3
  Week 156: number analyzed (Participants) | 114
  Week 156 | 97.4
  Week 172: number analyzed (Participants) | 187
  Week 172 | 98.4
  Week 188: number analyzed (Participants) | 62
  Week 188 | 100
  Week 204: number analyzed (Participants) | 99
  Week 204 | 94.9
  Week 220: number analyzed (Participants) | 138
  Week 220 | 97.8
  Week 236: number analyzed (Participants) | 10
  Week 236 | 100
  End of Study (Extension): number analyzed (Participants) | 324
  End of Study (Extension) | 96.9

12. Secondary Outcome: Percentage of Participants With EASI-90 (≥90% Reduction in EASI Scores From Baseline of the Parent Study) at Each Visit
Description: EASI-90 was defined as >=90% reduction in EASI scores from baseline of the parent study
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Week 4: number analyzed (Participants) | 2620
  Week 4 | 38.6
  Week 16: number analyzed (Participants) | 2560
  Week 16 | 57.7
  Week 36: number analyzed (Participants) | 1289
  Week 36 | 59.7
  Week 52: number analyzed (Participants) | 883
  Week 52 | 68.4
  Week 100: number analyzed (Participants) | 999
  Week 100 | 73.0
  Week 124: number analyzed (Participants) | 473
  Week 124 | 74.4
  Week 156: number analyzed (Participants) | 114
  Week 156 | 76.3
  Week 172: number analyzed (Participants) | 187
  Week 172 | 81.8
  Week 188: number analyzed (Participants) | 62
  Week 188 | 72.6
  Week 204: number analyzed (Participants) | 99
  Week 204 | 75.8
  Week 220: number analyzed (Participants) | 138
  Week 220 | 84.1
  Week 236: number analyzed (Participants) | 10
  Week 236 | 70.0
  End of Study (Extension): number analyzed (Participants) | 324
  End of Study (Extension) | 76.2

13. Secondary Outcome: Change From Baseline in Pruritus Numerical Rating Scale (NRS) in Parent Study
Description: The Pruritus NRS is an assessment tool for patients to report the intensity of their pruritus (itch), using a scale from 0-10, where 0 is no itch and 10 is the worst itch imaginable.
  Daily peak pruritus NRS score is the worst one between morning and evening scores of the day. Baseline Pruritus NRS is determined based on average of daily peak NRS scores during the 7 days immediately preceding randomization. A minimum of 4 daily scores out of 7 days is required to calculate baseline average score.
  Weekly worst score is calculated by taking the worst score within the week
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 1, 4, 16, 36, 52, 100, 124, 156, 172, 188, 204, 220, 236, 252, 272 (End of Study)"
Population: The safety analysis set (SAF) includes all patients who received any study drug; it is based on the treatment received. Participants recorded Pruritus score using IVRS (Interactive Voice Recording System) at specified timepoints
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Score on a Scale
  Week 1: number analyzed (Participants) | 2150
  Week 1 | -2.86 (2.492)
  Week 4: number analyzed (Participants) | 2249
  Week 4 | -3.81 (2.403)
  Week 16: number analyzed (Participants) | 1865
  Week 16 | -4.44 (2.377)
  Week 36: number analyzed (Participants) | 1924
  Week 36 | -4.67 (2.365)
  Week 52: number analyzed (Participants) | 1579
  Week 52 | -4.76 (2.371)
  Week 100: number analyzed (Participants) | 875
  Week 100 | -4.69 (2.315)
  Week 124: number analyzed (Participants) | 590
  Week 124 | -4.56 (2.359)
  Week 156: number analyzed (Participants) | 391
  Week 156 | -4.37 (2.352)
  Week 172: number analyzed (Participants) | 291
  Week 172 | -4.64 (2.256)
  Week 188: number analyzed (Participants) | 241
  Week 188 | -4.73 (2.194)
  Week 204: number analyzed (Participants) | 200
  Week 204 | -4.83 (2.341)
  Week 220: number analyzed (Participants) | 192
  Week 220 | -4.90 (2.231)
  Week 236: number analyzed (Participants) | 189
  Week 236 | -4.81 (2.308)
  Week 252: number analyzed (Participants) | 178
  Week 252 | -4.89 (2.201)
  Week 272: number analyzed (Participants) | 135
  Week 272 | -4.69 (2.238)

14. Secondary Outcome: Percent Change From Baseline in Pruritus NRS
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percent Change
  Week 1: number analyzed (Participants) | 1846
  Week 1 | -9.55 (40.989)
  Week 4: number analyzed (Participants) | 1859
  Week 4 | -28.88 (41.792)
  Week 16: number analyzed (Participants) | 1520
  Week 16 | -38.96 (47.891)
  Week 36: number analyzed (Participants) | 1595
  Week 36 | -41.38 (52.300)
  Week 52: number analyzed (Participants) | 1316
  Week 52 | -46.41 (41.912)
  Week 100: number analyzed (Participants) | 708
  Week 100 | -50.62 (42.112)
  Week 124: number analyzed (Participants) | 454
  Week 124 | -51.47 (39.063)
  Week 156: number analyzed (Participants) | 297
  Week 156 | -48.16 (55.076)
  Week 172: number analyzed (Participants) | 247
  Week 172 | -50.30 (42.907)
  Week 188: number analyzed (Participants) | 191
  Week 188 | -50.56 (43.444)
  Week 204: number analyzed (Participants) | 169
  Week 204 | -52.53 (43.465)
  Week 220: number analyzed (Participants) | 162
  Week 220 | -51.18 (39.244)
  Week 236: number analyzed (Participants) | 160
  Week 236 | -51.67 (37.690)
  Week 252: number analyzed (Participants) | 148
  Week 252 | -51.01 (47.328)
  Week 272: number analyzed (Participants) | 111
  Week 272 | -46.23 (46.404)

15. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Pruritus NRS ≥3 From Baseline
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Week 1: number analyzed (Participants) | 2204
  Week 1 | 11.9
  Week 4: number analyzed (Participants) | 2304
  Week 4 | 28.3
  Week 16: number analyzed (Participants) | 1908
  Week 16 | 39.3
  Week 36: number analyzed (Participants) | 1969
  Week 36 | 43.8
  Week 52: number analyzed (Participants) | 1609
  Week 52 | 45.9
  Week 100: number analyzed (Participants) | 893
  Week 100 | 51.1
  Week 124: number analyzed (Participants) | 601
  Week 124 | 48.8
  Week 156: number analyzed (Participants) | 396
  Week 156 | 46.5
  Week 172: number analyzed (Participants) | 294
  Week 172 | 54.1
  Week 188: number analyzed (Participants) | 242
  Week 188 | 52.5
  Week 204: number analyzed (Participants) | 202
  Week 204 | 56.9
  Week 220: number analyzed (Participants) | 194
  Week 220 | 51.5
  Week 236: number analyzed (Participants) | 191
  Week 236 | 51.3
  Week 252: number analyzed (Participants) | 178
  Week 252 | 56.2
  Week 272: number analyzed (Participants) | 136
  Week 272 | 50.0

16. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Pruritus NRS ≥4 From Baseline
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants
  Week 1: number analyzed (Participants) | 2204
  Week 1 | 7.0
  Week 4: number analyzed (Participants) | 2304
  Week 4 | 18.6
  Week 16: number analyzed (Participants) | 1908
  Week 16 | 29.3
  Week 36: number analyzed (Participants) | 1969
  Week 36 | 33.3
  Week 52: number analyzed (Participants) | 1609
  Week 52 | 35.4
  Week 100: number analyzed (Participants) | 893
  Week 100 | 41.4
  Week 124: number analyzed (Participants) | 601
  Week 124 | 39.4
  Week 156: number analyzed (Participants) | 396
  Week 156 | 35.6
  Week 172: number analyzed (Participants) | 294
  Week 172 | 42.9
  Week 188: number analyzed (Participants) | 242
  Week 188 | 40.9
  Week 204: number analyzed (Participants) | 202
  Week 204 | 44.1
  Week 220: number analyzed (Participants) | 194
  Week 220 | 40.2
  Week 236: number analyzed (Participants) | 191
  Week 236 | 37.2
  Week 252: number analyzed (Participants) | 178
  Week 252 | 42.7
  Week 272: number analyzed (Participants) | 136
  Week 272 | 36.0

17. Secondary Outcome: Percentage of Participants Requiring Rescue Treatment: Overall
Time Frame: Up to 272 weeks
Population: This included all participants who received any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants | 1.7

18. Secondary Outcome: Percentage of Participants Requiring Rescue Treatment: Systemic Treatment
Time Frame: Up to 272 weeks
Population: This included all participants who received any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants | 1.6

19. Secondary Outcome: Percentage of Participants Requiring Rescue Treatment: Phototherapy
Time Frame: Up to 272 weeks
Population: This included all participants who received any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Percentage of Participants | 0.0747

20. Secondary Outcome: Changes From Current Study Baseline to Prespecified Time Points Through the End of the Study: Dermatology Life Quality Index (DLQI)
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The format is a simple response to 10 items, which assess QOL over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor QOL
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 12, 24, 36, 48, 76, 100, 124, 148, 272 (End of Study)"
Population: Administered only to the subset of participants who fluently spoke the language for which a validated translation of the questionnaire was available, at time points according to the Schedule of Events as described in the study protocol. This included all participants who received any study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Score on a scale
  Baseline of Current Study | 8.5 (7.11)
  Week 12: number analyzed (Participants) | 2200
  Week 12 | -4.9 (5.93)
  Week 24: number analyzed (Participants) | 1601
  Week 24 | -6.0 (6.41)
  Week 36: number analyzed (Participants) | 1300
  Week 36 | -6.5 (6.51)
  Week 48: number analyzed (Participants) | 2243
  Week 48 | -5.6 (6.20)
  Week 76: number analyzed (Participants) | 415
  Week 76 | -7.2 (6.41)
  Week 100: number analyzed (Participants) | 877
  Week 100 | -7.3 (6.66)
  Week 124: number analyzed (Participants) | 118
  Week 124 | -7.9 (6.40)
  Week 148: number analyzed (Participants) | 11
  Week 148 | -8.3 (5.14)
  End of Study: number analyzed (Participants) | 69
  End of Study | -3.6 (7.37)

21. Secondary Outcome: Changes From Current Study Baseline to Prespecified Time Points Through the End of the Study: Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults. The format is a response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) with a scoring system of 0 to 28; a high score is indicative of a poor QOL.
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 12, 24, 36, 48, 76, 100, 124, 148, 272 (End of Study)"
Population: Administered only to the subset of participants who fluently speak the language for which a validated translation of the questionnaire is available. This included all participants who received any study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Score on a scale
  Week 12: number analyzed (Participants) | 2205
  Week 12 | -7.7 (7.32)
  Week 24: number analyzed (Participants) | 1598
  Week 24 | -9.3 (7.44)
  Week 36: number analyzed (Participants) | 1302
  Week 36 | -10.0 (7.46)
  Week 48: number analyzed (Participants) | 2247
  Week 48 | -8.8 (7.46)
  Week 76: number analyzed (Participants) | 422
  Week 76 | -11.6 (7.79)
  Week 100: number analyzed (Participants) | 879
  Week 100 | -11.4 (7.30)
  Week 124: number analyzed (Participants) | 118
  Week 124 | -12.7 (7.11)
  Week 148: number analyzed (Participants) | 11
  Week 148 | -10.5 (6.06)
  End of Study: number analyzed (Participants) | 70
  End of Study | -4.5 (10.91)

22. Secondary Outcome: Changes From Parent Study Baseline to Prespecified Time Points Through the End of the Study: EuroQol-5D (EQ-5D)
Description: The EuroQOL 5-Dimension Health Questionnaire (EQ-5D) is a standardized measure of health status developed by the EuroQOL Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The minimum value for the single index utility score is -0.594 (Best imaginable health state) and the maximum value for the single index utility score is 1 (Worst imaginable health state).
Time Frame: Up to 272 weeks (End of Study), "Baseline, Weeks 12, 24, 36, 48, 76, 100, 124, 148, 272 (End of Study)"
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 2677
Score on a scale
  Week 12: number analyzed (Participants) | 1909
  Week 12 | 0.2769 (0.31571)
  Week 24: number analyzed (Participants) | 1327
  Week 24 | 0.3001 (0.32062)
  Week 36: number analyzed (Participants) | 1047
  Week 36 | 0.3056 (0.33204)
  Week 48: number analyzed (Participants) | 1994
  Week 48 | 0.2854 (0.31017)
  Week 76: number analyzed (Participants) | 314
  Week 76 | 0.2965 (0.30658)
  Week 100: number analyzed (Participants) | 752
  Week 100 | 0.3217 (0.33832)
  Week 124: number analyzed (Participants) | 95
  Week 124 | 0.3242 (0.28937)
  Week 148: number analyzed (Participants) | 7
  Week 148 | 0.3046 (0.26337)
  End of Study: number analyzed (Participants) | 52
  End of Study | 0.1864 (0.32838)

23. Secondary Outcome: OPTIONAL SUB-STUDY: Ctrough of Functional Dupilumab in Serum Before and After Switching to the New Dupilumab Drug Product
Time Frame: Up to week 12
Population: The sub-study ADA population includes all treated patients who receive new dupilumab drug product and have at least one non-missing anti-dupilumab antibody result at any time during the sub-study period after the first dose of new dupilumab drug product.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab
Number analyzed (Participants) | 50
mg/L
  Week 0 | 65.9 (40.8)
  Week 12: number analyzed (Participants) | 48
  Week 12 | 65.4 (34.7)

24. Secondary Outcome: OPTIONAL SUB-STUDY: Incidence of Treatment-emergent Anti-drug Antibody (ADA) Response in Patients Receiving the New Dupilumab Drug Product
Description: For participants receiving dupilumab from a new manufacturing process, ADA baseline was defined as the baseline visit in the sub-study, or at the end of the main study, dependent on available data.
Time Frame: Up to 24 Weeks
Population: The sub-study ADA population includes all treated patients who receive new dupilumab drug product and have at least one non-missing anti-dupilumab antibody result at any time during the sub-study period after the first dose of new dupilumab drug product. No data collected.
Arm/Group | Dupilumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose to end of study (plus extension), approximately 272 weeks
Description: Participants received repeated doses of dupilumab
Arm/Group | Dupilumab
All-Cause Mortality (participants affected / at risk) | 3/2677
Serious Adverse Events (participants affected / at risk) | 283/2677
Other Adverse Events (participants affected / at risk) | 1613/2677
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=2677)
Appendicitis (Infections and infestations) | 6 (6)
Corona virus infection (Infections and infestations) | 3 (3)
Erysipelas (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3)
Pilonidal cyst (Infections and infestations) | 3 (3)
Chronic tonsillitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (3)
Eczema herpeticum (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Keratitis bacterial (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Superinfection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral corneal ulcer (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (14)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Granular cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease lymphocyte predominance type stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (12)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 5 (6)
Migraine (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 5 (5)
Colitis (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (2)
Cataract (Eye disorders) | 3 (3)
Ectropion (Eye disorders) | 2 (2)
Entropion (Eye disorders) | 2 (2)
Trichiasis (Eye disorders) | 2 (2)
Atopic keratoconjunctivitis (Eye disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Corneal erosion (Eye disorders) | 1 (3)
Corneal neovascularisation (Eye disorders) | 1 (2)
Corneal perforation (Eye disorders) | 1 (1)
Eyelid cyst (Eye disorders) | 1 (1)
Keratoconus (Eye disorders) | 1 (1)
Mydriasis (Eye disorders) | 1 (1)
Optic neuropathy (Eye disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (7)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Chordae tendinae rupture (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Panic attack (Psychiatric disorders) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
"Schizophrenia, paranoid type" (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (5)
Calculus ureteric (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Death (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (3)
Chest pain (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 3 (4)
Food allergy (Immune system disorders) | 2 (2)
Contrast media allergy (Immune system disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Congenital knee deformity (Congenital, familial and genetic disorders) | 1 (1)
Dolichocolon (Congenital, familial and genetic disorders) | 1 (1)
Goitre (Endocrine disorders) | 2 (2)
Thyroid mass (Endocrine disorders) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Female sterilisation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=2677)
Nasopharyngitis (Infections and infestations) | 774 (1602)
Upper respiratory tract infection (Infections and infestations) | 365 (567)
Conjunctivitis (Infections and infestations) | 277 (417)
Oral herpes (Infections and infestations) | 200 (463)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 446 (787)
Conjunctivitis allergic (Eye disorders) | 242 (329)
Headache (Nervous system disorders) | 218 (411)
Injection site reaction (General disorders) | 138 (506)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT01949311/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT01949311/SAP_001.pdf